CLINICAL TRIAL: NCT04368156
Title: A Prospective, Randomized, Controlled Study Assessing Vagus Nerve Stimulation in CoViD-19 Respiratory Symptoms (SAVIOR)
Brief Title: Study Assessing Vagus Nerve Stimulation in CoViD-19 Respiratory Symptoms
Acronym: SAVIOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carlos Tornero (Other)
Responsible Party: Sponsor-Investigator, Carlos Tornero, Doctor, Hospital Clínico Universitario de Valencia
Organization: Hospital Clínico Universitario de Valencia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAVIOR
Record Dates: First submitted 2020-04-20; First posted 2020-04-29 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19 | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (No Intervention)
- Gammacore treatment (Experimental)
  Interventions: Device: gammaCore® (Vagus nerve stimulation)

INTERVENTIONS:
Device: gammaCore® (Vagus nerve stimulation) — Vagus nerve stimulation using the gammacore neurostimulation device
  Arms: Gammacore treatment

SUMMARY:
The purpose of this study is to asses the efficacy of the Gammacore device reducing the need for mechanical ventilation in patients diagnosed of Covid-19

ELIGIBILITY:
Inclusion Criteria:

1. Has been tested positive or suspected/presumed positive for CoViD-19
2. Patients with cough, shortness of breath or respiratory compromise (RR>24/min, increased work of breathing.)
3. O2 Saturation less than or equal to 96% on room air or sensation
4. Agrees to use the gammaCore®-Sapphire device as intended and to follow all of the requirements of the study including recording required study data
5. Patient is able to provide signed and witnessed Informed Consent

Exclusion Criteria:

1. On home/therapy oxygen (i.e. for COPD patients) at baseline prior to development of CoViD-19
2. Is already enrolled in a clinical trial using immunotherapeutic regimen for CoViD-19
3. Already gammaCore for other medical conditions
4. A history of aneurysm, intracranial hemorrhage, brain tumors, or significant head trauma
5. Known or suspected severe atherosclerotic cardiovascular disease, severe carotid artery disease (eg, bruits or history of transient ischemic attack or cerebrovascular accident), congestive heart failure, known severe coronary artery disease, or recent myocardial infarction
6. Uncontrolled high blood pressure (>140/90)
7. Current implantation of an electrical and/or neurostimulator device, including but not limited to a cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant
8. Current implantation of metal cervical spine hardware or a metallic implant near the gammaCore stimulation site
9. Belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with the follow-up requirements, or provide self-assessments is compromised (e.g. homeless, developmentally disabled and prisoner)
10. Compromised access to peripheral veinous for blood)
11. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Incidence of changes in specific clinical events in patients with covid-19. | From randomization to hospital discharge or ICU admission, whatever occurs first, assessed up to two months
  The clinical events include, but are not limited, to:
  * Proportion of subjects requiring mechanical ventilation
  * Days to onset of mechanical ventilation
  * Oxygen support requirements
  * O2 saturation
  * Pain levels
  * PaO2/FiO2
  * Coagulation
  * Laboratory measurements related to circulating cytokines and inflammation.
  * Live discharge from the hospital
  * Patient length of stay
  * Mortality
  * Need for intensive care
  * Shortness of breath
  * Device related serious adverse events
  * Adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1 Staats, P., et al. (2018). In E.Krames, et. al (Eds.) Neuromodulation : Comprehensive Textbook of Principles, Technologies, and Therapies Vol 1: Neurostiumulation for Asthma (2nd Edition, pp. 1339-1345). London, United Kingdom: Academic Press, Elsevier.
- [Background] Miner JR, Lewis LM, Mosnaim GS, Varon J, Theodoro D, Hoffmann TJ. Feasibility of percutaneous vagus nerve stimulation for the treatment of acute asthma exacerbations. Acad Emerg Med. 2012 Apr;19(4):421-9. doi: 10.1111/j.1553-2712.2012.01329.x. PMID 22506946
- [Background] Pavlov VA, Chavan SS, Tracey KJ. Bioelectronic Medicine: From Preclinical Studies on the Inflammatory Reflex to New Approaches in Disease Diagnosis and Treatment. Cold Spring Harb Perspect Med. 2020 Mar 2;10(3):a034140. doi: 10.1101/cshperspect.a034140. PMID 31138538
- [Background] Hoffmann TJ, Mendez S, Staats P, Emala CW, Guo P. Inhibition of histamine-induced bronchoconstriction in Guinea pig and Swine by pulsed electrical vagus nerve stimulation. Neuromodulation. 2009 Oct;12(4):261-9. doi: 10.1111/j.1525-1403.2009.00234.x. Epub 2009 Aug 20. PMID 22151415
- [Background] Koopman FA, Chavan SS, Miljko S, Grazio S, Sokolovic S, Schuurman PR, Mehta AD, Levine YA, Faltys M, Zitnik R, Tracey KJ, Tak PP. Vagus nerve stimulation inhibits cytokine production and attenuates disease severity in rheumatoid arthritis. Proc Natl Acad Sci U S A. 2016 Jul 19;113(29):8284-9. doi: 10.1073/pnas.1605635113. Epub 2016 Jul 5. PMID 27382171
- [Background] Brock C, Brock B, Aziz Q, Moller HJ, Pfeiffer Jensen M, Drewes AM, Farmer AD. Transcutaneous cervical vagal nerve stimulation modulates cardiac vagal tone and tumor necrosis factor-alpha. Neurogastroenterol Motil. 2017 May;29(5). doi: 10.1111/nmo.12999. Epub 2016 Dec 12. PMID 27957782
- [Background] Tarn J, Legg S, Mitchell S, Simon B, Ng WF. The Effects of Noninvasive Vagus Nerve Stimulation on Fatigue and Immune Responses in Patients With Primary Sjogren's Syndrome. Neuromodulation. 2019 Jul;22(5):580-585. doi: 10.1111/ner.12879. Epub 2018 Oct 17. PMID 30328647
- [Background] Lerman I, Hauger R, Sorkin L, Proudfoot J, Davis B, Huang A, Lam K, Simon B, Baker DG. Noninvasive Transcutaneous Vagus Nerve Stimulation Decreases Whole Blood Culture-Derived Cytokines and Chemokines: A Randomized, Blinded, Healthy Control Pilot Trial. Neuromodulation. 2016 Apr;19(3):283-90. doi: 10.1111/ner.12398. Epub 2016 Mar 15. PMID 26990318
- [Background] Huston JM, Gallowitsch-Puerta M, Ochani M, Ochani K, Yuan R, Rosas-Ballina M, Ashok M, Goldstein RS, Chavan S, Pavlov VA, Metz CN, Yang H, Czura CJ, Wang H, Tracey KJ. Transcutaneous vagus nerve stimulation reduces serum high mobility group box 1 levels and improves survival in murine sepsis. Crit Care Med. 2007 Dec;35(12):2762-8. doi: 10.1097/01.CCM.0000288102.15975.BA. PMID 17901837
- [Background] Haveri A, Smura T, Kuivanen S, Osterlund P, Hepojoki J, Ikonen N, Pitkapaasi M, Blomqvist S, Ronkko E, Kantele A, Strandin T, Kallio-Kokko H, Mannonen L, Lappalainen M, Broas M, Jiang M, Siira L, Salminen M, Puumalainen T, Sane J, Melin M, Vapalahti O, Savolainen-Kopra C. Serological and molecular findings during SARS-CoV-2 infection: the first case study in Finland, January to February 2020. Euro Surveill. 2020 Mar;25(11):2000266. doi: 10.2807/1560-7917.ES.2020.25.11.2000266. PMID 32209163
- [Background] Conti P, Ronconi G, Caraffa A, Gallenga CE, Ross R, Frydas I, Kritas SK. Induction of pro-inflammatory cytokines (IL-1 and IL-6) and lung inflammation by Coronavirus-19 (COVI-19 or SARS-CoV-2): anti-inflammatory strategies. J Biol Regul Homeost Agents. 2020 March-April,;34(2):327-331. doi: 10.23812/CONTI-E. PMID 32171193
- [Background] Liu L, Wei Q, Lin Q, Fang J, Wang H, Kwok H, Tang H, Nishiura K, Peng J, Tan Z, Wu T, Cheung KW, Chan KH, Alvarez X, Qin C, Lackner A, Perlman S, Yuen KY, Chen Z. Anti-spike IgG causes severe acute lung injury by skewing macrophage responses during acute SARS-CoV infection. JCI Insight. 2019 Feb 21;4(4):e123158. doi: 10.1172/jci.insight.123158. eCollection 2019 Feb 21. PMID 30830861
- [Background] Chen IY, Moriyama M, Chang MF, Ichinohe T. Severe Acute Respiratory Syndrome Coronavirus Viroporin 3a Activates the NLRP3 Inflammasome. Front Microbiol. 2019 Jan 29;10:50. doi: 10.3389/fmicb.2019.00050. eCollection 2019. PMID 30761102
- [Background] Gralinski LE, Sheahan TP, Morrison TE, Menachery VD, Jensen K, Leist SR, Whitmore A, Heise MT, Baric RS. Complement Activation Contributes to Severe Acute Respiratory Syndrome Coronavirus Pathogenesis. mBio. 2018 Oct 9;9(5):e01753-18. doi: 10.1128/mBio.01753-18. PMID 30301856
- [Background] McDermott JE, Mitchell HD, Gralinski LE, Eisfeld AJ, Josset L, Bankhead A 3rd, Neumann G, Tilton SC, Schafer A, Li C, Fan S, McWeeney S, Baric RS, Katze MG, Waters KM. The effect of inhibition of PP1 and TNFalpha signaling on pathogenesis of SARS coronavirus. BMC Syst Biol. 2016 Sep 23;10(1):93. doi: 10.1186/s12918-016-0336-6. PMID 27663205
- [Background] Newton AH, Cardani A, Braciale TJ. The host immune response in respiratory virus infection: balancing virus clearance and immunopathology. Semin Immunopathol. 2016 Jul;38(4):471-82. doi: 10.1007/s00281-016-0558-0. Epub 2016 Mar 10. PMID 26965109
- [Background] Gralinski LE, Ferris MT, Aylor DL, Whitmore AC, Green R, Frieman MB, Deming D, Menachery VD, Miller DR, Buus RJ, Bell TA, Churchill GA, Threadgill DW, Katze MG, McMillan L, Valdar W, Heise MT, Pardo-Manuel de Villena F, Baric RS. Genome Wide Identification of SARS-CoV Susceptibility Loci Using the Collaborative Cross. PLoS Genet. 2015 Oct 9;11(10):e1005504. doi: 10.1371/journal.pgen.1005504. eCollection 2015 Oct. PMID 26452100
- [Background] Selinger C, Tisoncik-Go J, Menachery VD, Agnihothram S, Law GL, Chang J, Kelly SM, Sova P, Baric RS, Katze MG. Cytokine systems approach demonstrates differences in innate and pro-inflammatory host responses between genetically distinct MERS-CoV isolates. BMC Genomics. 2014 Dec 22;15(1):1161. doi: 10.1186/1471-2164-15-1161. PMID 25534508
- [Background] Burrack KS, Morrison TE. The role of myeloid cell activation and arginine metabolism in the pathogenesis of virus-induced diseases. Front Immunol. 2014 Sep 8;5:428. doi: 10.3389/fimmu.2014.00428. eCollection 2014. PMID 25250029
- [Background] van den Brand JM, Haagmans BL, van Riel D, Osterhaus AD, Kuiken T. The pathology and pathogenesis of experimental severe acute respiratory syndrome and influenza in animal models. J Comp Pathol. 2014 Jul;151(1):83-112. doi: 10.1016/j.jcpa.2014.01.004. Epub 2014 Jan 15. PMID 24581932
- [Background] DeDiego ML, Nieto-Torres JL, Regla-Nava JA, Jimenez-Guardeno JM, Fernandez-Delgado R, Fett C, Castano-Rodriguez C, Perlman S, Enjuanes L. Inhibition of NF-kappaB-mediated inflammation in severe acute respiratory syndrome coronavirus-infected mice increases survival. J Virol. 2014 Jan;88(2):913-24. doi: 10.1128/JVI.02576-13. Epub 2013 Nov 6. PMID 24198408
- [Background] Smits SL, de Lang A, van den Brand JM, Leijten LM, van IJcken WF, Eijkemans MJ, van Amerongen G, Kuiken T, Andeweg AC, Osterhaus AD, Haagmans BL. Exacerbated innate host response to SARS-CoV in aged non-human primates. PLoS Pathog. 2010 Feb 5;6(2):e1000756. doi: 10.1371/journal.ppat.1000756. PMID 20140198
- [Background] Kong SL, Chui P, Lim B, Salto-Tellez M. Elucidating the molecular physiopathology of acute respiratory distress syndrome in severe acute respiratory syndrome patients. Virus Res. 2009 Nov;145(2):260-9. doi: 10.1016/j.virusres.2009.07.014. Epub 2009 Jul 25. PMID 19635508
- [Background] Wan J, Sun W, Li X, Ying W, Dai J, Kuai X, Wei H, Gao X, Zhu Y, Jiang Y, Qian X, He F. Inflammation inhibitors were remarkably up-regulated in plasma of severe acute respiratory syndrome patients at progressive phase. Proteomics. 2006 May;6(9):2886-94. doi: 10.1002/pmic.200500638. PMID 16649161
- [Background] Okabayashi T, Kariwa H, Yokota S, Iki S, Indoh T, Yokosawa N, Takashima I, Tsutsumi H, Fujii N. Cytokine regulation in SARS coronavirus infection compared to other respiratory virus infections. J Med Virol. 2006 Apr;78(4):417-24. doi: 10.1002/jmv.20556. PMID 16482545
- [Background] Yu SY, Hu YW, Liu XY, Xiong W, Zhou ZT, Yuan ZH. Gene expression profiles in peripheral blood mononuclear cells of SARS patients. World J Gastroenterol. 2005 Aug 28;11(32):5037-43. doi: 10.3748/wjg.v11.i32.5037. PMID 16124062
- [Background] Yang YH, Huang YH, Chuang YH, Peng CM, Wang LC, Lin YT, Chiang BL. Autoantibodies against human epithelial cells and endothelial cells after severe acute respiratory syndrome (SARS)-associated coronavirus infection. J Med Virol. 2005 Sep;77(1):1-7. doi: 10.1002/jmv.20407. PMID 16032747
- [Background] Wang CH, Liu CY, Wan YL, Chou CL, Huang KH, Lin HC, Lin SM, Lin TY, Chung KF, Kuo HP. Persistence of lung inflammation and lung cytokines with high-resolution CT abnormalities during recovery from SARS. Respir Res. 2005 May 11;6(1):42. doi: 10.1186/1465-9921-6-42. PMID 15888207
- [Background] Steyn E, Mohamed Z, Husselman C. Non-invasive vagus nerve stimulation for the treatment of acute asthma exacerbations-results from an initial case series. Int J Emerg Med. 2013 Mar 19;6(1):7. doi: 10.1186/1865-1380-6-7. PMID 23510361
- [Background] Tisoncik JR, Korth MJ, Simmons CP, Farrar J, Martin TR, Katze MG. Into the eye of the cytokine storm. Microbiol Mol Biol Rev. 2012 Mar;76(1):16-32. doi: 10.1128/MMBR.05015-11. PMID 22390970
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Background] Mourdoukoutas AP, Truong DQ, Adair DK, Simon BJ, Bikson M. High-Resolution Multi-Scale Computational Model for Non-Invasive Cervical Vagus Nerve Stimulation. Neuromodulation. 2018 Apr;21(3):261-268. doi: 10.1111/ner.12706. Epub 2017 Oct 27. PMID 29076212
- [Background] Henssen DJHA, Derks B, van Doorn M, Verhoogt N, Van Cappellen van Walsum AM, Staats P, Vissers K. Vagus nerve stimulation for primary headache disorders: An anatomical review to explain a clinical phenomenon. Cephalalgia. 2019 Aug;39(9):1180-1194. doi: 10.1177/0333102419833076. Epub 2019 Feb 20. PMID 30786731
- [Background] Fornai F, Ruffoli R, Giorgi FS, Paparelli A. The role of locus coeruleus in the antiepileptic activity induced by vagus nerve stimulation. Eur J Neurosci. 2011 Jun;33(12):2169-78. doi: 10.1111/j.1460-9568.2011.07707.x. Epub 2011 May 3. PMID 21535457
- [Derived] Tornero C, Pastor E, Garzando MDM, Orduna J, Forner MJ, Bocigas I, Cedeno DL, Vallejo R, McClure CK, Czura CJ, Liebler EJ, Staats P. Non-invasive Vagus Nerve Stimulation for COVID-19: Results From a Randomized Controlled Trial (SAVIOR I). Front Neurol. 2022 Apr 8;13:820864. doi: 10.3389/fneur.2022.820864. eCollection 2022. PMID 35463130
- [Derived] Tornero C, Vallejo R, Cedeno D, Orduna J, Pastor E, Belaouchi M, Escamilla B, Laredo M, Del Mar Garzando M. A prospective, randomized, controlled study assessing vagus nerve stimulation using the gammaCore(R)-Sapphire device for patients with moderate to severe CoViD-19 Respiratory Symptoms (SAVIOR): A structured summary of a study protocol for a randomised controlled trial". Trials. 2020 Jun 26;21(1):576. doi: 10.1186/s13063-020-04486-w. PMID 32586395